CLINICAL TRIAL: NCT06533033
Title: Melatonin Epigenetic Potential in Preventing Malignant Transformation of Oral Lichen Planus Epigenetic Randomized Clinical Trial
Brief Title: Melatonin Epigenetic Potential in Preventing Malignant Transformation of Oral Lichen Planus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Clinical invesitgator and Biostatistical consultanat, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Melatonin_2023
Record Dates: First submitted 2024-07-25; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- melatonin therapy (Experimental)
  Interventions: Drug: Rapid Release Capsules Melatoni
- topical corticosteroid a (Active Comparator)
  Interventions: Drug: Triamcinolone Acetonide ointment, Kenacort-A orabase

INTERVENTIONS:
Drug: Rapid Release Capsules Melatoni — Twenty-five will be given melatonin therapy in combination with the conventional treatment.
  2 tablets,30 minutes before sleeping once daily for 8 weeks.
  Arms: melatonin therapy
Drug: Triamcinolone Acetonide ointment, Kenacort-A orabase — Twenty-five will be given topical corticosteroid applied twice to three times daily.
  Topical antifungal will be applied three to four times daily. This conventional treatment will be given to the patients for 8 weeks
  Arms: topical corticosteroid a

SUMMARY:
Background: Oral Lichen planus (OLP) is one of the most common oral diseases that has an unneglectable rate of malignant transformation. Recently malignant transformation has been definitively linked to epigenetic changes. One of those most common changes is DNA hypermethylation that causes tumor suppressor genes to downtranslate and thus carcinogenesis begins. ZNF582 gene hypermethylation is emerging as an exclusive biomarker to differentiate between normal and dysplastic changes that occur over the epithelium. Aim: To evaluate the Melatonin epigenetic potential in preventing malignant transformation of OLP. Material and methods: an epigenetic randomized clinical study will be conducted on 50 patients suffering from OLP, recruited from the outpatient clinic of Oral medicine department, Alexandria Faculty of Dentistry, Egypt. Patients will be assigned to either Control group who will receive topical corticosteroids and antifungal treatment, or test group who will receive melatonin supplement in addition to conventional treatment. All patients will be genetically evaluated for the level of DNA hypermethylation 8 weeks after treatment, and clinically evaluated for disease severity and pain, by Elsabagh scoring system 4. 8, and 12 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically and histopathologically diagnosed to be suffering from OLP in the following forms has been reported in the literature to have the highest potentiality for malignant transformation (plaque-type lichen , Erosive lichen planus, ulcerative lichen planus), with or without histopathological dysplasia.
* Patients who have symptoms (i.e. pain and burning sensation) secondary to OLP.

Exclusion Criteria:

* Patients suspected to have lichenoid drug reaction or lichenoid contact allergy.
* Patients suffering from systemic diseases (such as diabetes, cardiovascular or liver disorders, renal dysfunction).
* Patients with findings of any physical or mental abnormality that would interfere with or be affected by the study procedure.
* Patients who have adverse habits of chewing tobacco and smoking.
* Pregnant and lactating women.
* Patients under treatment with corticosteroids and immunosuppressants.
* Patients exhibiting any skin manifestations of OLP

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
change in DNA methylation level of tumor suppressor gene (ZNF852) | up to 8 weeks
  The ZNF582 gene sequence will be obtained from the University of California, Santa Cruz, Genomics Institute.
  website (http://genome.ucsc.edu/), and the methylation-specific PCR primers for ZNF582 will be acquired from MethPrimer (http://www.urogene.org/cgibin/ methprimer/methprimer.cgi).
Change in oral lesions | Up to 12 weeks
  Oral lesions will be evaluated clinically after treatment using Elsabagh et al score.
  Objective mucosal lesion nature (no lesion= 0, White keratotic lesion =1, Atrophy/Erosion intermixed or not with White lesion = 2, Ulceration intermixed or not with White lesion = 3)
Change in pain scores | Up to 12 weeks
  Subjective pain score (no pain =0, mild pain=1, moderate pain=2, severe pain=3)
Change in number of affected surfaces in oral cavity | Up to 12 weeks
  Number of surfaces affected in the oral cavity other than the gingiva (only one surface affected or buccal mucosae bilaterally =0, more than one surface affected or more than both buccal mucosae=1)
Change in gingival involvement | Up to 12 weeks
  Gingival involvement as desquamative gingivitis (no gingival involvement = 0, narrow band (1mm) of gingival involvement or wide band in less than 6 teeth involved =1, wide band (>1mm) of gingival involvement in more than 6 teeth involved = 2)

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral medicine Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Egypt